CLINICAL TRIAL: NCT03790735
Title: Targeted Chromosomal Aberrations Detection by FISH Analysis of Circulating Abnormal Cells to Differentiate of Benign and Malignant Pulmonary Nodules
Brief Title: The MDA Test to Differentiate of Benign and Malignant Pulmonary Nodules
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Zhuhai livzon cynvenio diagnostics LTD (Unknown)
Responsible Party: Sponsor
Other Study IDs: TianjinCIH2018
Record Dates: First submitted 2018-12-28; First posted 2019-01-02 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Pulmonary Nodule, Solitary
Keywords: pulmonary nodule
MeSH Terms: conditions — Solitary Pulmonary Nodule

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diagnostic test: Targeted chromosomal aberrations detection by FISH (MDA TEST).
  Interventions: Diagnostic Test: FISH

INTERVENTIONS:
Diagnostic Test: FISH — Targeted chromosomal aberrations detection

SUMMARY:
* The purpose of the study is the identification of the efficacy of MDA Test to Differentiate of Benign and Malignant Pulmonary Nodules.
* In this study, the investigators are going to validate the efficacy of the MDA test for diagnosing early lung cancer by comparing results of the pre-surgery MDA test with the post-surgery pathology.

DETAILED DESCRIPTION:
* Current state-of-the-art lung cancer early screening utilizes low-dose CT scan to identify lung nodules smaller than 3 cm in diameter. However, it's still a clinical challenge to differentiate between malignant and benign nodules.
* This study is being conducted to evaluate the efficacy of the MDA TEST to detect Targeted chromosomal aberrations in circulating abnormal cells by FISH analysis that might be an early indicator of lung cancer. Approximately 200 Pre-surgery adult patients with single pulmonary nodule found by CT scan, will be enrolled in the study. The sample type of MDA test is Peripheral Blood. This study will compare the results of the pre-surgery MDA Test with the post-surgery pathology to determine if the test can detect lung cancer or the lack of lung cancer .
* The results of the test will not be provided to the subject, the investigator and will not be used to diagnose or treat the subject.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or above
* single pulmonary nodule found by CT scan.
* the diameter of the pulmonary nodule is between 5mm to 30mm.
* plan to accept pneumonectomy due to the pulmonary nodule.
* agree to sign informed consent

Exclusion Criteria:

* fail to understand or agree to sign informed consent.
* pregnant or lactating women.
* the diameter of the pulmonary nodule is more than 30mm.
* there are 2 or more pulmonary nodules in one single patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 200 participants
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-05-03 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Early detection of lung cancer | 6 months
  The efficacy of the MDA TEST assay comparing with pathologic diagnosis(the gold standard), and CT/LDCT diagnosis, including sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV).

CONTACTS AND LOCATIONS:
Overall Officials: Changli Wang, Prof, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute & Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: Undecided